CLINICAL TRIAL: NCT07190287
Title: Evaluation of a Wearable EEG-tFUS System for REM Sleep Modulation in Healthy Adults and Individuals With Subclinical Sleep Disturbances
Brief Title: Wearable Neural Interfacing System for REM Sleep Restoration and Enhancement
Acronym: NEUSleeP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Evan (Huiliang) Wang, Assistant Professor, University of Texas at Austin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005703; HR00112490328 (Other Grant/Funding Number: DEFENSE ADVANCED RESEARCH PROJECTS AGENCY)
Record Dates: First submitted 2025-07-31; First posted 2025-09-24 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Sleep Disturbance; Stress, Psychological; REM Sleep Measurement
Keywords: Transcranial Focused Ultrasound (tFUS); Wearable EEG; Sleep Modulation; REM Sleep; Subthalamic Nucleus; Closed-Loop Neuromodulation; Non-invasive Brain Stimulation; Stress Adaptation; Neural Interface
MeSH Terms: conditions — Parasomnias; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Two cohorts in parallel: (1) Healthy adults and (2) adults with subclinical sleep/stress disturbance. Each participant completes two consecutive overnight visits-Night 1 baseline (no stimulation) and Night 2 tFUS with EEG-guided REM-timed delivery-enabling within-subject comparisons (baseline vs stimulation) in each cohort. An imaging-validation subset of healthy volunteers completes a same-day MRI-FUS session with pre/post fMRI to verify targeting and neural engagement. Operational "phases" (device checks, imaging validation, healthy sleep study, subclinical sleep study) are procedural and do not imply staged allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Healthy Volunteers - NEUSleeP Validation and Modulation (Experimental): Participants will undergo three phases: (1) NEUSleeP device validation through biweekly EEG and impedance testing over 4 weeks (subset of participants); (2) STN targeting validation using BrainSonix and NEUSleeP with structural MRI and fMRI to assess BOLD response in the STN; and (3) overnight REM sleep modulation with NEUSleeP including EEG/EMG/EOG recordings and pre/post fMRI scans to assess stress-related brain activity and REM sleep outcomes.
  Interventions: Device: NEUSleeP system (FUS-EEG wearable device); Device: BrainSonix Pulsar 1002
- Subclinical Sleep Disturbance Group - NEUSleeP REM Modulation (Experimental): Participants with non-clinical sleep and stress disturbances (PSQI 5-10, PSS 16-21) will undergo baseline overnight EEG/EMG/EOG recording followed by a second night of NEUSleeP-guided FUS stimulation targeting the STN. Pre- and post-intervention fMRI scans and stress questionnaires will assess neural and behavioral effects.
  Interventions: Device: NEUSleeP system (FUS-EEG wearable device)

INTERVENTIONS:
Device: NEUSleeP system (FUS-EEG wearable device) — The NEUSleeP system is a wearable FUS-EEG device integrating hydrogel-based EEG and focused ultrasound neuromodulation. The intervention includes:
  1. Device testing in 4 healthy volunteers to assess EEG signal and impedance over 4 weeks vs. wet electrodes;
  2. STN targeting validation in up to 20 participants using MRI-guided tFUS with NEUSleeP and BrainSonix Pulsar 1002, with fMRI analysis of BOLD activation in stress-related areas (amygdala, insula);
  3. REM sleep modulation in 16 healthy participants across two nights, evaluating REM sleep architecture and stress-related fMRI changes following STN stimulation during REM;
  4. A similar protocol in 12 individuals with self-reported poor sleep and moderate stress, assessing subjective stress (PSS), sleep dynamics, and connectivity changes post-tFUS.
Device: BrainSonix Pulsar 1002 — The BrainSonix Pulsar 1002 is a research-grade focused ultrasound device used to evaluate STN targeting in up to 20 healthy participants. COMSOL 2D acoustic simulations and structural MRI are used to localize the STN. The BrainSonix system is tuned and installed for STN stimulation during fMRI scanning. Pre- and post-stimulation fMRI is conducted to verify BOLD signal changes in the STN and related regions. These responses are compared with those from NEUSleeP stimulation, using identical imaging protocols. Ultrasound parameters are iteratively adjusted to optimize targeting while adhering to FDA diagnostic ultrasound safety limits. A linear mixed model is used to assess stimulation-induced changes.
  Arms: Healthy Volunteers - NEUSleeP Validation and Modulation

SUMMARY:
This study evaluates a wearable system (NEUSleeP) that combines overnight EEG recording with transcranial focused ultrasound (tFUS) targeted to deep brain structures involved in REM sleep regulation (e.g., subthalamic nucleus). The primary objective is to assess safety and estimate effects on REM sleep quantity and architecture; secondary objectives include changes in stress-related measures.

Healthy adults aged 18-50, with or without subclinical sleep or stress complaints, will complete two consecutive overnight recordings: Night 1 (baseline, no stimulation) and Night 2 (tFUS, EEG-guided and timed to REM). Participants will complete stress questionnaires. fMRI is conducted using two paradigms: in an imaging-validation subset, pre- and post-stimulation scans are acquired in the same MRI-FUS session; in the two-night cohorts, scans are acquired the morning before and the morning after the FUS night to assess BOLD responses.

Outcomes include REM time, REM percentage, number of REM periods, REM latency, safety/tolerability, and exploratory neuroimaging and self-reported stress measures. Findings will inform the feasibility of a wearable EEG-tFUS approach to modulate REM sleep and stress adaptation.

DETAILED DESCRIPTION:
This study evaluates the safety, feasibility, and preliminary signals of effect of NEUSleeP, a wearable neural interface for closed-loop modulation of REM sleep using transcranial focused ultrasound (tFUS) targeted to the subthalamic nucleus (STN). The system integrates a flexible ultrasound transducer with bioadhesive hydrogel EEG electrodes in a patch designed for repeated overnight use. REM sleep is implicated in emotional regulation, memory processes, and stress adaptation. Existing noninvasive approaches have focused largely on NREM modulation; this study examines a REM-focused, target-directed approach to determine whether tFUS delivered during sleep can alter REM architecture and related outcomes.

The study comprises four phases:

Phase 1 (device functionality) enrolls four healthy volunteers for repeated bench and on-body checks (EEG signal quality, contact impedance stability, usability) over four weeks, with comparisons to standard clinical electrodes.

Phase 2 (STN stimulation and imaging validation) uses structural MRI and acoustic modeling to configure STN targeting for both a reference research system (BrainSonix Pulsar 1002) and NEUSleeP. In up to 20 healthy volunteers, functional MRI is acquired immediately before and immediately after the same MRI-FUS session to characterize BOLD responses in STN and stress-related networks (e.g., amygdala, insula), using identical imaging protocols across platforms.

Phase 3 (REM modulation in healthy volunteers) enrolls 16 adults for two consecutive overnight recordings: Night 1 baseline (no stimulation) and Night 2 tFUS (closed-loop stimulation time-locked to REM using EEG). Primary sleep outcomes include REM time, REM percentage, number of REM periods, and REM latency; safety and tolerability are recorded throughout.

Phase 4 (REM modulation in participants with non-clinical sleep disturbance) enrolls 12 adults with elevated sleep complaints and perceived stress for the same two-night protocol; exploratory outcomes include self-reported stress measures collected around the FUS night.

Two fMRI paradigms are used across phases. In Phase 2, a same-session MRI-FUS visit includes pre-stimulation and post-stimulation fMRI acquisitions in the same session (healthy imaging-validation subset). In Phases 3 and 4, participants complete morning-before (pre-FUS night) and morning-after (post-FUS night) fMRI sessions to assess changes around the overnight REM-timed stimulation.

Safety procedures include MRI screening where applicable, continuous adverse event capture, stop rules for stimulation, and post-visit follow-up. Ultrasound exposure is controlled within established diagnostic ultrasound limits (e.g., MI <= 1.9 and derated time-averaged intensity within applicable FDA limits), with device-level acoustic verification prior to use. Data monitoring is performed by the study team with predefined criteria for pausing or discontinuation. Findings will inform the feasibility of a wearable EEG-tFUS approach for REM-related modulation and guide parameters for future controlled trials.

ELIGIBILITY:
Inclusion Criteria for Healthy Volunteers:

- Adults aged 18-50, willing and able to undergo MRI, EEG, and FUS experiments.

Inclusion Criteria for Healthy Volunteers with Non-Clinical Sleep Disturbances:

* Adults aged 18-50, willing and able to undergo EEG and FUS experiments.
* Pittsburgh Sleep Quality Index (PSQI) score between 5 and 10.
* Perceived Stress Scale (PSS) score between 16 and 21.

Exclusion Criteria for Both Groups:

* Current or past history of psychopathology, epilepsy, or other seizure disorders.
* Inability to provide informed consent to undergo EEG recording, FUS stimulation, and MRI.
* Diagnosed sleep disorders (e.g., insomnia, obstructive sleep apnea).
* Contraindications to FUS or MRI, including but not limited to: history of stroke, brain tumors, brain hemorrhages, internal wires, electrodes, pacemakers, implants, irremovable ferromagnetic objects in the head that are unsafe for MRI and/or cause large imaging artifacts, brain surgery, moderate-to-severe head injury, any penetrating head injury, or uncontrolled thyroid disorder.
* Pregnant individuals or those attempting to become pregnant (due to unknown MRI-related risks to fetuses).
* Serious medical illnesses likely to interfere with study participation.
* Current active suicidal or homicidal ideation (or suicide attempt within the past 3 months).
* Current substance use disorder.
* Current or recent (within the past 3 months) psychotic symptoms.
* Currently meeting diagnostic criteria for a manic episode.
* Currently engaged in evidence-based or experimental treatments (e.g., weekly cognitive behavioral therapy, transcranial magnetic stimulation, ketamine/esketamine treatment) other than psychiatric medications that have been on a stable dosage and regimen for at least 3 months (including antidepressants, mood stabilizers, atypical antipsychotics, and sedatives/hypnotics), in order to avoid confounding therapeutic effects.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Total REM Sleep Time | Night 1 (Baseline) and Night 2 (FUS); consecutive nights.
  This measure evaluates the difference in total time (minutes) spent in rapid eye movement (REM) sleep between the baseline and stimulation nights, as recorded via EEG during overnight polysomnography. The goal is to assess whether STN-targeted tFUS delivered by NEUSLeeP enhances REM sleep duration.
Change in REM Sleep Percentage of Total Sleep Time | Night 1 (Baseline) and Night 2 (FUS); consecutive nights.
  Percentage of total sleep time spent in REM sleep will be compared between the baseline and stimulation nights to determine whether NEUSLeeP tFUS enhances REM architecture.
Change in STN BOLD Signal Following Ultrasound Stimulation | pre-FUS (≤15 minutes before) and post-FUS (≤15 minutes after).
  This outcome measures the change in blood-oxygen-level-dependent (BOLD) signal in the subthalamic nucleus (STN) before and after transcranial focused ultrasound (tFUS) stimulation using NEUSleeP and BrainSonix devices. Functional MRI will be used to assess activation in the STN and related regions (e.g., amygdala, insula). The goal is to evaluate device efficacy in modulating STN activity.

SECONDARY OUTCOMES:
Change in Number of REM Sleep Cycles | Night 1 (Baseline) and Night 2 (FUS); consecutive nights.
  The number of distinct REM sleep cycles will be recorded on both baseline and stimulation nights to evaluate the effect of STN-targeted tFUS on REM cycling.
Change in REM Sleep Latency | Night 1 (Baseline) and Night 2 (FUS); consecutive nights.
  Time (in minutes) from sleep onset to the first REM episode will be measured and compared between the baseline and stimulation nights to assess whether tFUS shortens REM latency.
Change in Subjective Stress Levels (PSQ Score) | Night 2 (FUS): pre (≤24 hours before) and post (≤24 hours after).
  Participants will complete the Perceived Stress Questionnaire (PSQ) before and after the stimulation night. Changes in PSQ scores will assess the effect of STN-targeted tFUS on perceived stress.
Change in Stress-Related Brain Connectivity and Activation (fMRI) | Day 2 morning (pre-FUS night) and Day 3 morning (post-FUS night).
  Resting-state BOLD fMRI will assess changes in amygdala and insula connectivity before and after the stimulation night. In addition, an fMRI facial emotion recognition task will evaluate activation changes in stress-related neural circuits.

CONTACTS AND LOCATIONS:
Overall Officials: Huiliang (Evan) Wang, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- UT Austin, Biomedical Engineering Department, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Summers J, Nowicki M. Managing organizational improvement in a resource-challenged environment. Healthc Financ Manage. 2002 Jul;56(7):60-2. No abstract available. PMID 12119832
- [Background] Cicolin A, Lopiano L, Zibetti M, Torre E, Tavella A, Guastamacchia G, Terreni A, Makrydakis G, Fattori E, Lanotte MM, Bergamasco B, Mutani R. Effects of deep brain stimulation of the subthalamic nucleus on sleep architecture in parkinsonian patients. Sleep Med. 2004 Mar;5(2):207-10. doi: 10.1016/j.sleep.2003.10.010. PMID 15033145
- [Background] Legon W, Sato TF, Opitz A, Mueller J, Barbour A, Williams A, Tyler WJ. Transcranial focused ultrasound modulates the activity of primary somatosensory cortex in humans. Nat Neurosci. 2014 Feb;17(2):322-9. doi: 10.1038/nn.3620. Epub 2014 Jan 12. PMID 24413698